CLINICAL TRIAL: NCT06443749
Title: Closure of the Appendiceal Stump With a Polymer Clip Versus Intracorporeal Ligation With a Single Instrument in Laparoscopic Appendectomy; Prospective Randomized Trial
Brief Title: Closure of the Appendiceal Stump
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sezgin Topuz (Other)
Responsible Party: Sponsor-Investigator, Sezgin Topuz, assistant professor, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAHRAMANMARASKSUGCSTOPUZ1.....
Record Dates: First submitted 2023-12-11; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Appendectomy
Keywords: Appendectomy
MeSH Terms: interventions — Appendectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group1 (Active Comparator): the appendiceal stump will be closed with a polyper homologous clip
  Interventions: Procedure: appendectomy
- group (Active Comparator): the stump will be closed with an intracorporial node with a single instrument in
  Interventions: Procedure: appendectomy

INTERVENTIONS:
Procedure: appendectomy — the appendiceal stump will be closed with a polyper homologous clip or with an intracorporial node

SUMMARY:
Laparoscopic appendectomy is a well-defined surgical technique. However, concerns remain about whether closure of the appendiceal stump should be done with clips, endoloops, staples, or other techniques. If tying is to be used in the closure of the appendiceal stump, there is no consensus on which technique (intracorporoyal, extracorporoyal, etc.) should be used for ligation. For this reason, there is a need for studies on different binding techniques and instruments currently used. The aim of this study was to compare the use of unilateral intracorporeal knot and polymer endoclip closure during laparoscopic appendectomy.

DETAILED DESCRIPTION:
Patients who are scheduled to undergo laparoscopic appendectomy after the ethics committee approval will be included consecutively. Patients will be randomized into 2 groups: those who will be closed with a polymer endoclip (Group 1) and those who will be closed with an intracorporeal node with a single instrument (Group 2). Data such as age, gender, body mass index, comorbidities, previous abdominal surgeries, medications used by the patients, as well as the presence of ileus, perforation, and diffuse peritonitis will be recorded. After laparoscopic dissection, the appendiceal stump will be closed with a polyper homologous clip in Group 1 and the stump will be closed with an intracorporial node with a single instrument in Group 2. The operation times of the patients, the time elapsed after the end of the dissection until the pathology specimen comes out of the skin (to be determined as the closure time), complications such as ileus, intra-abdominal abscess, bleeding and fistula related to stump closure problems encountered in the postoperative period will be recorded and compared. Patients will be followed by the corresponding author In both surgical methods, it is routinely used to close the appendiceal stump and in the polymer clip application, a clip with a locking mechanism is used when the stump is tightened with an applicator. In the intracorporial node with one hand, the surgical node is made by circulating the tip of the suture material around the appendix with a single instrument (the other end is kept fixed outside the abdomen)

ELIGIBILITY:
Inclusion Criteria

* Patients who are diagnosed with acute appendicitis

Exclusion Criteria:

* bleeding diathesis
* cirrhotic acid,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
operation time | 3 months
  operation time

IPD SHARING:
Plan to Share IPD: No